CLINICAL TRIAL: NCT05522257
Title: Expression of Prostate Specific Membrane Antigen (PSMA) in Soft Tissue Sarcomas and Urothelial Cell Carcinomas: Implications for Tumour-specific Molecular Imaging and Treatment?
Brief Title: PSMA Expression and PSMA PET Imaging in Soft Tissue Sarcomas and Urothelial Cell Carcinomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Lioe-Fee de Geus-Oei, MD PhD, Prof. dr. L.F. de Geus-Oei, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL78279.058.21
Record Dates: First submitted 2022-08-16; First posted 2022-08-31 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Sarcoma,Soft Tissue; Urothelial Carcinoma
Keywords: Prostate Specific Membrane Antigen; Soft Tissue Sarcoma; Urothelial Carcinoma; Urothelial Neoplasm; Transitional Cell Carcinoma; PSMA; PSMA PET/CT; JK-PSMA-7
MeSH Terms: conditions — Sarcoma; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: This pilot study is a single centre, open-label, phase II study in patients with advanced soft tissue sarcoma (cohort 1) and advanced urothelial cell carcinoma (cohort 2). It is a non-randomized, non-blinded, prospective pilot study to assess the level of PSMA expression and the feasibility of PSMA-targeted theranostics in these patient groups. In all patients that are included in this pilot study, immunohistochemical PSMA staining will be performed on their biopsy material. In case of high PSMA expression, as defined by previous literature, a [18F]-JK-PSMA-7 PET/CT scan will be made to assess the level of tracer uptake in the malignant lesion(s). The expected duration of recruitment is 1 year and 9 months. An early stopping rule of 5 negative PSMA PET/CT scans is implemented in this study, for each cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Advanced soft tissue sarcoma (n=60) and advanced urothelial cell carcinoma (n=60) (Other): The study population comprises sixty adult patients with diagnosis of advanced (locally irresectable or metastasized) soft tissue sarcoma (cohort 1) and sixty adult patients with diagnosis of advanced (muscle invasive or metastasized) urothelial cell carcinoma (cohort 2).
  Interventions: Diagnostic Test: [18F]-JK-PSMA-7 PET/CT scan

INTERVENTIONS:
Diagnostic Test: [18F]-JK-PSMA-7 PET/CT scan — A [18F]-JK-PSMA-7 PET/CT scan will be made to assess the level of tracer uptake in the malignant lesion(s). We expect to make a [18F]-JK-PSMA-7 PET/CT scan in 15 out of 60 patients per cohort.

SUMMARY:
This pilot study aims to investigate the PSMA expression in the biopsy material of advanced soft tissue sarcomas and advanced urothelial cell carcinomas, and in case of high PSMA expression (as defined by previous literature), to investigate whether this correlates with high tracer uptake on PSMA-targeted PET. This way, (a subset of) patients can be selected that could benefit from radionuclide targeted therapy in the future.

DETAILED DESCRIPTION:
Background:

Patients with metastatic soft tissue sarcoma and metastatic urothelial cell carcinoma have a poor prognosis, with a five-year survival rate of 16% and 6%, respectively. This is due to limited treatment options and low response rates to systemic chemotherapy of approximately 25% in soft tissue sarcomas and 40-50% in urothelial cell carcinomas. In these patient groups there is a high need for new effective treatment options that can decrease burden of disease and increase survival benefit.

Prostate specific membrane antigen (PSMA) is a transmembrane metallopeptidase that is overexpressed in prostate cancer cells. For diagnostic purposes, PET/CT scans that target PSMA have found their way into the clinical routine of prostate cancer patients. However, currently we know that despite the name, PSMA is not prostate cancer specific. It is also found in the tumour-associated blood vessels of a wide variety of other tumours, including soft tissue sarcomas and urothelial cell carcinomas. In many different sarcoma types, PSMA expression is seen in the neovasculature with the highest detection rate of 46-60% in high grade and undifferentiated sarcomas (e.g. pleomorphic sarcoma types). The PSMA expression rate in the neovasculature of urothelial cell carcinomas still varies in literature, however, the most recently published article showed that PSMA expression was found in 93% of urothelial cell carcinoma tissues. Additionally, PSMA expression was seen in the tumour cells itself in 79% of the tissues. Because of the unique expression pattern which seems to be limited to tumour cells and tumour-associated endothelial cells, PSMA may represent an interesting target for molecular imaging using PSMA-targeting PET scans, and eventually for radionuclide targeted therapy, when coupled to an alpha- or beta-emitter. [225Act]-PSMA and [177Lu]-PSMA therapy have shown promising results in the treatment of advanced prostate cancer patients and might offer perspective and increase quality of life in patients with advanced soft tissue sarcoma and urothelial cell carcinoma, as well.

Objective of the study:

This pilot study aims to investigate the PSMA expression in the biopsy material of advanced soft tissue sarcomas and advanced urothelial cell carcinomas, and in case of high PSMA expression (as defined by previous literature), to investigate whether this correlates with high tracer uptake on PSMA-targeted PET. This way, (a subset of) patients can be selected that could benefit from radionuclide targeted therapy in the future.

Study design:

This pilot study is a single centre, open-label, non-randomized, non-blinded phase II study with two patient cohorts.

Study population:

The study population comprises sixty adult patients with diagnosis of advanced (locally irresectable or metastasized) soft tissue sarcoma (cohort 1) and sixty adult patients with diagnosis of advanced (muscle invasive or metastasized) urothelial cell carcinoma (cohort 2). The expected duration of recruitment is 1 year and 9 months.

Intervention:

In all included patients, biopsy material is obtained as part of routine clinical practice. For this study, immunohistochemical PSMA staining will be performed on these biopsy materials. If the biopsy material shows high PSMA expression (as defined by previous literature), a [18F]-JK-PSMA-7 PET/CT scan will be made to assess the level of tracer uptake in the malignant lesion(s). We expect to make a [18F]-JK-PSMA-7 PET/CT scan in 15 out of 60 patients in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years at the time of informed consent.
* Diagnosis of advanced (locally irresectable or metastasized) soft tissue sarcoma (cohort 1) or advanced (muscle invasive or metastasized) urothelial cell carcinoma (cohort 2).
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.
* Recent (< 8 weeks) standard imaging (with CT or [18F]-FDG PET/CT) with measurable disease (lesion diameter > 1 cm).
* Biopsy available of primary tumour and/or metastasis
* WHO performance status of 0-2
* Either:

  * No previous systemic therapy for advanced soft tissue sarcoma or advanced urothelial cell carcinoma, or;
  * Previous systemic therapy for advanced soft tissue sarcoma or advanced urothelial cell carcinoma with progression of disease during systemic therapy or progression of disease after discontinuation of systemic therapy, or;
  * Previous systemic therapy for advanced soft tissue sarcoma or advanced urothelial cell carcinoma with partial response or stable disease, where the last dose of systemic therapy was given > 8 weeks before.

Exclusion Criteria:

* Women who are pregnant and/or lactating.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Known hypersensitivity to drugs comparative to [18F]-JK-PSMA-7, any of their excipients or to any component of [18F]-JK-PSMA-7.
* Inability to undergo PET/CT scanning, e.g. claustrophobia, weight limits or inability to tolerate lying down for the duration of a PET/CT scan (~30 minutes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Quantify PSMA-tracer accumulation and determine whether SUV > 8 | 6 months
  To quantify the accumulation of [18F]-JK-PSMA-7 on PET/CT imaging by using the standardized uptake values (SUV) and to determine the number of patients in which the SUVmax in advanced soft tissue sarcoma (cohort 1) and advanced urothelial cell carcinoma (cohort 2) is higher than 8. In these patients, PSMA-targeted radioligand therapy might be beneficial in the future.

SECONDARY OUTCOMES:
Correlation between PSMA expression and PSMA-tracer uptake | 6 months
  Assessing if higher levels of PSMA expression in biopsy material result in higher levels of PSMA-tracer uptake on a [18F]-JK-PSMA-7 PET/CT scan.
Correlation PSMA expression and tumour grade, tumour stage and tumour subtype | 6 months
  The correlation between PSMA expression in biopsy material and tumour grade, tumour stage (TNM system) and histological subtype, as concluded by the pathologist.
Histological differences between primary tumours and metastases | 6 months
  The immunohistochemical PSMA expression pattern in primary tumours vs. metastases
Differences on [18F]-JK-PSMA-7 PET/CT between primary tumours and metastases | 6 months
  Quantified PSMA-tracer uptake (SUVmax) in primary tumours vs. metastases
Agreement between [18F]-JK-PSMA-7 PET/CT and standard imaging | 6 months
  The number of detected lesions on [18F]-JK-PSMA-7 PET/CT vs. standard imaging (CT or [18F]-FDG PET/CT)

CONTACTS AND LOCATIONS:
Overall Officials: Lioe-Fee De Geus-Oei, prof.dr., Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Patient data includes medical history and imaging data, which cannot be completely anonymized.

REFERENCES:
- [Derived] Kleiburg F, van der Hulle T, Gelderblom H, Slingerland M, Speetjens FM, Hawinkels LJAC, Dibbets-Schneider P, van Velden FHP, Pool M, Lam SW, Bovee JVMG, Heijmen L, de Geus-Oei LF. PSMA expression and PSMA PET/CT imaging in metastatic soft tissue sarcoma patients, results of a prospective study. Eur J Nucl Med Mol Imaging. 2025 Aug;52(10):3690-3699. doi: 10.1007/s00259-025-07224-z. Epub 2025 Mar 27. PMID 40146266